CLINICAL TRIAL: NCT06906107
Title: Validation of a Clinical Prediction Rule to Identify Patients With Neck Pain Likely to Benefit From Cervical Spinal Manipulation: A Randomized Clinical Trial
Brief Title: Validating a Clinical Prediction Rule to Guide Manual Therapy and Exercise for Neck Pain Relief in 140 Participants With Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: Foundation for Physical Therapy Research (Other)
Responsible Party: Principal Investigator, Jessica Feda, Clinical Assistant Professor, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2240854-1
Record Dates: First submitted 2025-03-18; First posted 2025-04-02 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain Musculoskeletal; Neck Pain Treatment; Cervicalgia
Keywords: neck pain; manual therapy; physical therapy
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The initial investigator performing the baseline assessment is masked to the treatment. The investigator performing the treatment is masked to the initial investigator's assessment of the patient's categorization on the clinical prediction rule. The outcome assessor is masked to the intervention received and status on the clinical prediction rule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Manipulation (Experimental): Patients will receive cervical manipulation on 2 visits, followed by 3 visits of therapeutic exercise.
  Interventions: Procedure: Cervical Manipulation; Procedure: Exercise
- Exercise and Mobilizations (Other): Patients will receive low-grade cervical mobilizations on 2 visits, followed by 3 visits of therapeutic exercises
  Interventions: Procedure: Exercise; Procedure: Mobilization

INTERVENTIONS:
Procedure: Cervical Manipulation — High velocity low amplitude thrust joint manipulation to the cervical spine facet joints
  Arms: Cervical Manipulation
Procedure: Exercise — Therapeutic exercises to the cervical, thoracic, and scapular musculature
Procedure: Mobilization — Low velocity, low amplitude movements applied to the cervical spine facet joints (Grade I or II)
  Arms: Exercise and Mobilizations

SUMMARY:
Neck pain is a common issue that can lead to long-term disability and lost work time for many individuals. Despite numerous studies, finding effective treatment strategies has been challenging. One possible reason for this is that treatments may not have been tested on the specific groups of people who would benefit most. A method was developed to identify people with neck pain who are likely to see significant improvements from a manipulation technique used by physical therapists, called cervical spine thrust joint manipulation. The investigators believe that patients identified as likely responders to cervical spine manipulation will show greater improvements in disability. The investigators aim to test whether this method works with different patients and therapists across the country through a multicenter randomized clinical trial. In this study, 140 patients with primary complaints of neck pain will be enrolled from 20 clinical sites. Designed with stringent criteria for inclusion, this study is a testament to our commitment to participant safety and the effectiveness of the treatment. Participants will be randomly assigned to one of two groups: (1) one group will receive 2 sessions of cervical spine manipulation followed by 3 sessions of exercise, and (2) the other group will receive 2 sessions of gentle hands-on treatment followed by 3 sessions of exercise. The primary goal is to measure changes in disability 4 weeks after starting treatment, with follow-ups after one week, 4 weeks, 3 months, and 6 months to assess both immediate and long-term effects. By providing crucial data on the reliability of our method in identifying patients who will benefit most from cervical spine manipulation, this study has the potential to significantly enhance decision-making leading to rapid improvement. Results from this study will provide clearer guidelines on the optimal use of cervical spine manipulation, potentially revolutionizing the way patients recover from neck pain.

DETAILED DESCRIPTION:
This study's primary objective will examine whether a previously derived clinical prediction rule (CPR) exhibits validity for identifying a subgroup of patients who respond favorably to cervical thrust joint manipulation (C-TJM). The secondary objective will determine if patients who are positive on the derived CPR and receive C-TJM will exhibit reduced downstream healthcare costs. This multicenter randomized clinical trial will enroll 140 patients with primary complaints of neck pain. Participants will be randomized into two groups: (1) 2 sessions of C-TJM followed by 3 sessions of stretching and strengthening exercises, and (2) 2 sessions of low-grade mobilizations followed by 3 sessions of the same stretching and strengthening exercises. The primary outcome is the change in disability measured four weeks post-treatment, with pain as the secondary outcome. Follow-up assessments will occur at one week, 4 weeks, 3 months and 6 months to evaluate both short-term and long-term effects. The exact inclusion and exclusion criteria from the CPR derivation study will be used within this validation study to determine participant eligibility. Data will be collected using standardized self-report measures and physical examination, and statistical analyses will be performed using a linear mixed model with repeated measures. The investigators hypothesize that patients identified by the clinical prediction rule to benefit from C-TJM will show substantial improvements in disability and pain. This study will offer valuable insight into the effectiveness of C-TJM for neck pain. Successful validation of the clinical prediction rule could lead to more efficient and cost-effective patient care, potentially reducing the burden of neck pain on healthcare systems and improving patient outcomes. As PI, responsibilities include protocol development, training, data collection, analysis, manuscript development and dissemination of findings.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 70
* Primary complaint of neck pain with or without unilateral upper extremity symptoms
* Neck Disability Index (NDI) score of 10 or greater
* Numeric Pain Rating Scale score of 2 or greater

Exclusion Criteria:

* History of whiplash injury within the past 6 weeks
* Diagnosis of cervical spinal stenosis
* Bilateral upper extremity symptoms
* Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumor, fracture, rheumatoid arthritis, osteoporosis, severe atherosclerosis, dizziness, diplopia, drop attacks, bilateral numbness, nausea, prolonged history of steroid use)
* Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes)
* Two or more positive neurological signs consistent with significant nerve root compression, including any two of the following:

  1. Muscle weakness involving a major muscle group of the upper extremity
  2. Diminished upper extremity muscle stretch reflex (biceps, triceps, or brachioradialis)
  3. Diminished or absent sensation to pinprick or light touch in any upper extremity dermatome
* Prior neck surgery
* Current pregnancy, pregnancy within 6 months, or currently lactating
* Pending legal action pertaining to their neck pain
* Inability to read English at the 8th grade reading level
* Inability to legally provide informed consent for any other reason
* Inability to comply with the treatment and follow-up schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 6 months
  10-item patient self-report measure of perceived disability. Each question is scored from 0 to 5. Minimum value of 0 and maximum value of 50. Higher scores indicate worse disability and a poorer outcome.

SECONDARY OUTCOMES:
Global Rating of Change Scale | 6 months
  A 15-point scale with options ranging from -7 (a great deal worse) to +7 (a great deal better) to determine the magnitude of change in response to intervention. Higher scores indicate a better outcome. Minimum value -7 and maximum value +7.
Numeric Pain Rating Scale | 6 months
  Patients rate their pain on a scale from 0 to 10, with 0 representing no pain and 10 representing the worst possible. Minimum value 0 and maximum value 10. Higher scores indicate a worse outcome.
Fear Avoidance Beliefs Questionnaire | 6 months
  A 16 question outcome measure scaled from 0 to 6 with a maximum score of 96 - a higher score indicates fear avoidance behaviors. Minimum score 0 and maximum score 96.
Medication Use | 6 months
  Self-report of medication use prior to, during, and after the treatment phase of the study. As this component is a self-report of medication use, scoring is not pertinent.
Healthcare Utilization | 6 months
  Self-report of healthcare use prior to and after the treatment phase of the study. As this component is a self-report of healthcare use, scoring is not pertinent.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica T Feda, DSc, Principal Investigator — Baylor University; Emilio J Puentedura, PhD, Study Director — Baylor University
Locations (3):
- United States (3):
  - ActivePT, Rochester, Minnesota
  - PROActivePT, Syracuse, New York
  - ActiveTherapy Alliance, Waco, Texas

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers beyond what will be published within future manuscripts and disseminations. However, if an individual researcher was to request IPD sharing upon completion of data analysis and dissemination, we would certainly consider the request.

REFERENCES:
- [Result] Childs JD, Fritz JM, Flynn TW, Irrgang JJ, Johnson KK, Majkowski GR, Delitto A. A clinical prediction rule to identify patients with low back pain most likely to benefit from spinal manipulation: a validation study. Ann Intern Med. 2004 Dec 21;141(12):920-8. doi: 10.7326/0003-4819-141-12-200412210-00008. PMID 15611489
- [Result] Cleland JA, Mintken PE, Carpenter K, Fritz JM, Glynn P, Whitman J, Childs JD. Examination of a clinical prediction rule to identify patients with neck pain likely to benefit from thoracic spine thrust manipulation and a general cervical range of motion exercise: multi-center randomized clinical trial. Phys Ther. 2010 Sep;90(9):1239-50. doi: 10.2522/ptj.20100123. Epub 2010 Jul 15. PMID 20634268
- [Result] Kaale BR, Krakenes J, Albrektsen G, Wester K. Clinical assessment techniques for detecting ligament and membrane injuries in the upper cervical spine region--a comparison with MRI results. Man Ther. 2008 Oct;13(5):397-403. doi: 10.1016/j.math.2007.03.007. Epub 2007 Nov 1. PMID 17936054
- [Result] Uitvlugt G, Indenbaum S. Clinical assessment of atlantoaxial instability using the Sharp-Purser test. Arthritis Rheum. 1988 Jul;31(7):918-22. doi: 10.1002/art.1780310715. PMID 3395385
- [Result] Hutting N, Scholten-Peeters GG, Vijverman V, Keesenberg MD, Verhagen AP. Diagnostic accuracy of upper cervical spine instability tests: a systematic review. Phys Ther. 2013 Dec;93(12):1686-95. doi: 10.2522/ptj.20130186. Epub 2013 Jul 25. PMID 23886844
- [Result] Hengeveld E, Banks K. Maitland's Vertebral Manipulation: Management of Neuromusculoskeletal Disorders - Volume 1. Elsevier Health Sciences; 2013.
- [Result] Piva SR, Erhard RE, Childs JD, Browder DA. Inter-tester reliability of passive intervertebral and active movements of the cervical spine. Man Ther. 2006 Nov;11(4):321-30. doi: 10.1016/j.math.2005.09.001. Epub 2006 Jul 11. PMID 16837235
- [Result] Harris KD, Heer DM, Roy TC, Santos DM, Whitman JM, Wainner RS. Reliability of a measurement of neck flexor muscle endurance. Phys Ther. 2005 Dec;85(12):1349-55. PMID 16305273
- [Result] Tong HC, Haig AJ, Yamakawa K. The Spurling test and cervical radiculopathy. Spine (Phila Pa 1976). 2002 Jan 15;27(2):156-9. doi: 10.1097/00007632-200201150-00007. PMID 11805661
- [Result] Wainner RS, Fritz JM, Irrgang JJ, Boninger ML, Delitto A, Allison S. Reliability and diagnostic accuracy of the clinical examination and patient self-report measures for cervical radiculopathy. Spine (Phila Pa 1976). 2003 Jan 1;28(1):52-62. doi: 10.1097/00007632-200301010-00014. PMID 12544957
- [Result] Cleland JA, Childs JD, Fritz JM, Whitman JM. Interrater reliability of the history and physical examination in patients with mechanical neck pain. Arch Phys Med Rehabil. 2006 Oct;87(10):1388-95. doi: 10.1016/j.apmr.2006.06.011. PMID 17023251
- [Result] Guidetti L, Placentino U, Baldari C. Reliability and Criterion Validity of the Smartphone Inclinometer Application to Quantify Cervical Spine Mobility. Clin Spine Surg. 2017 Dec;30(10):E1359-E1366. doi: 10.1097/BSD.0000000000000364. PMID 26905732
- [Result] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Result] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Result] Dunning JR, Cleland JA, Waldrop MA, Arnot CF, Young IA, Turner M, Sigurdsson G. Upper cervical and upper thoracic thrust manipulation versus nonthrust mobilization in patients with mechanical neck pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):5-18. doi: 10.2519/jospt.2012.3894. Epub 2011 Sep 30. PMID 21979312
- [Result] Cleland JA, Childs JD, Fritz JM, Whitman JM, Eberhart SL. Development of a clinical prediction rule for guiding treatment of a subgroup of patients with neck pain: use of thoracic spine manipulation, exercise, and patient education. Phys Ther. 2007 Jan;87(1):9-23. doi: 10.2522/ptj.20060155. Epub 2006 Dec 1. PMID 17142640
- [Result] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Result] Young BA, Walker MJ, Strunce JB, Boyles RE, Whitman JM, Childs JD. Responsiveness of the Neck Disability Index in patients with mechanical neck disorders. Spine J. 2009 Oct;9(10):802-8. doi: 10.1016/j.spinee.2009.06.002. Epub 2009 Jul 25. PMID 19632904
- [Result] Hoving JL, O'Leary EF, Niere KR, Green S, Buchbinder R. Validity of the neck disability index, Northwick Park neck pain questionnaire, and problem elicitation technique for measuring disability associated with whiplash-associated disorders. Pain. 2003 Apr;102(3):273-281. doi: 10.1016/S0304-3959(02)00406-2. PMID 12670669
- [Result] Jaeschke R, Singer J, Guyatt GH. A comparison of seven-point and visual analogue scales. Data from a randomized trial. Control Clin Trials. 1990 Feb;11(1):43-51. doi: 10.1016/0197-2456(90)90031-v. PMID 2157581
- [Result] Ritter PL, Gonzalez VM, Laurent DD, Lorig KR. Measurement of pain using the visual numeric scale. J Rheumatol. 2006 Mar;33(3):574-80. PMID 16511926
- [Result] Krebs EE, Carey TS, Weinberger M. Accuracy of the pain numeric rating scale as a screening test in primary care. J Gen Intern Med. 2007 Oct;22(10):1453-8. doi: 10.1007/s11606-007-0321-2. Epub 2007 Aug 1. PMID 17668269
- [Result] Fraenkel L, Falzer P, Fried T, Kohler M, Peters E, Kerns R, Leventhal H. Measuring pain impact versus pain severity using a numeric rating scale. J Gen Intern Med. 2012 May;27(5):555-60. doi: 10.1007/s11606-011-1926-z. Epub 2011 Nov 12. PMID 22081365
- [Result] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Result] Miyamoto GC, Lin CC, Cabral CMN, van Dongen JM, van Tulder MW. Cost-effectiveness of exercise therapy in the treatment of non-specific neck pain and low back pain: a systematic review with meta-analysis. Br J Sports Med. 2019 Feb;53(3):172-181. doi: 10.1136/bjsports-2017-098765. Epub 2018 Apr 20. PMID 29678893
- [Result] Toll DB, Janssen KJ, Vergouwe Y, Moons KG. Validation, updating and impact of clinical prediction rules: a review. J Clin Epidemiol. 2008 Nov;61(11):1085-94. doi: 10.1016/j.jclinepi.2008.04.008. PMID 19208371
- [Result] Childs JD, Cleland JA. Development and application of clinical prediction rules to improve decision making in physical therapist practice. Phys Ther. 2006 Jan;86(1):122-31. doi: 10.1093/ptj/86.1.122. No abstract available. PMID 16386067
- [Result] Puentedura EJ, Cleland JA, Landers MR, Mintken PE, Louw A, Fernandez-de-Las-Penas C. Development of a clinical prediction rule to identify patients with neck pain likely to benefit from thrust joint manipulation to the cervical spine. J Orthop Sports Phys Ther. 2012 Jul;42(7):577-92. doi: 10.2519/jospt.2012.4243. Epub 2012 May 14. PMID 22585595
- [Result] Kay TM, Gross A, Goldsmith CH, Rutherford S, Voth S, Hoving JL, Bronfort G, Santaguida PL. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD004250. doi: 10.1002/14651858.CD004250.pub4. PMID 22895940
- [Result] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Result] American Physical Therapy Association.. Guide to Physical Therapist Practice. Second Edition. American Physical Therapy Association. Phys Ther. 2001 Jan;81(1):9-746. No abstract available. PMID 11175682
- [Result] Dieleman JL, Cao J, Chapin A, Chen C, Li Z, Liu A, Horst C, Kaldjian A, Matyasz T, Scott KW, Bui AL, Campbell M, Duber HC, Dunn AC, Flaxman AD, Fitzmaurice C, Naghavi M, Sadat N, Shieh P, Squires E, Yeung K, Murray CJL. US Health Care Spending by Payer and Health Condition, 1996-2016. JAMA. 2020 Mar 3;323(9):863-884. doi: 10.1001/jama.2020.0734. PMID 32125402
- [Result] Safiri S, Kolahi AA, Hoy D, Buchbinder R, Mansournia MA, Bettampadi D, Ashrafi-Asgarabad A, Almasi-Hashiani A, Smith E, Sepidarkish M, Cross M, Qorbani M, Moradi-Lakeh M, Woolf AD, March L, Collins G, Ferreira ML. Global, regional, and national burden of neck pain in the general population, 1990-2017: systematic analysis of the Global Burden of Disease Study 2017. BMJ. 2020 Mar 26;368:m791. doi: 10.1136/bmj.m791. PMID 32217608
- [Result] GBD 2021 Neck Pain Collaborators. Global, regional, and national burden of neck pain, 1990-2020, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2024 Mar;6(3):e142-e155. doi: 10.1016/S2665-9913(23)00321-1. PMID 38383088
- [Result] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT06906107/Prot_SAP_ICF_000.pdf